CLINICAL TRIAL: NCT04141085
Title: Transcriptomic Evaluation of Endometrial Receptivity
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2019-01
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers without infertility: Healthy volunteers without a history of infertility who have regular menstrual cycles and whom have not had any intrauterine procedures performed in the last 90 days prior to participation in the study
  Interventions: Other: Endometrial biopsy
- Infertile Patients: Infertile patients with a history of infertility but without concern for endometrial dysfunction as the cause of their infertility.
  Interventions: Other: Endometrial biopsy

INTERVENTIONS:
Other: Endometrial biopsy — All groups will undergo a mock frozen embryo transfer cycle with an endometrial biopsy being performed as opposed to an embryo transfer

SUMMARY:
The purpose of this study is to comprehensively evaluate the transcriptomic signal of the endometrium before, during, and after the window of receptivity.

DETAILED DESCRIPTION:
Phase 1 will aim to define a normal endometrial transcriptomic signature in healthy controls without infertility. Phase 2 will elucidate endometrial transcriptomic expression in patients with diagnoses of infertility unrelated to endometrial factor. Findings from this phase will be compared to the results of phase 1.

ELIGIBILITY:
Phase 1:

Major Inclusion: The following are major inclusion criteria:

1. Regular menstrual cycles
2. Age 18-50
3. Normal baseline ultrasound
4. No intrauterine procedures in prior 90 days

Exclusions: The following are exclusion criteria:

1. Any contraindications to undergoing estrogen stimulation of the endometrium

   1. Current smoking status
   2. Multiple risk factors for arterial cardiovascular disease (smoking, diabetes, and hypertension)
   3. Hypertension (systolic ≥140 mmHg or diastolic ≥90 mmHg)
   4. Venous thromboembolism (current or history of)
   5. Known thrombogenic mutations
   6. Known ischemic heart disease
   7. History of stroke
   8. Complicated valvular heart disease (pulmonary hypertension, risk for atrial fibrillation, history of subacute bacterial endocarditis)
   9. Systemic lupus erythematosus (positive or unknown antiphospholipid antibodies)
   10. Migraine with aura at any age
   11. Breast cancer
   12. Cirrhosis
   13. Hepatocellular adenoma or malignant hepatoma
2. History of infertility diagnosis
3. History of undiagnosed abnormal uterine bleeding.
4. Allergic reaction to any medication used for the preparatory cycle
5. Known pregnancy or delivery within the past 6 months
6. Breastfeeding
7. Obesity >35 kg/m2

Phase 2

Major Inclusion: The following are major inclusion criteria:

1. Age 18-50
2. Diagnosis of infertility with low endometrial risk
3. No intrauterine procedures in prior 90 days

Exclusions: In addition to the exclusion criteria for phase 1, patients deemed to have an elevated endometrial risk will also be excluded. This would include the following:

1. Recurrent implantation failure
2. Failed transfer with a euploid blastocyst
3. History of Asherman's or abnormal endometrial function
4. History of endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Phase 1:
  Healthy volunteers without a history of infertility will be recruited for the first phase to undergo an endometrial biopsy on a randomized cycle day surrounding the window of implantation
  Phase 2:
  Healthy volunteers with a history of infertility but without concern for endometrial dysfunction will be recruited for the second phase to undergo an endometrial biopsy during a preparatory IVF cycle.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
transcriptomic evaluation | 90 days
  evaluation to characterize genes expressed during the window of implantation

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No